CLINICAL TRIAL: NCT02871505
Title: The Association Between Molecular Typing of Treponema Pallidum and Treatment Efficacy and Clinical Findings
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jun Li, Principal Investigator, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PUMCH-2016079
Record Dates: First submitted 2016-08-09; First posted 2016-08-18 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Syphilis
MeSH Terms: conditions — Syphilis | interventions — Penicillin G

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Molecular subtyping (14d/f) of Treponema pallidum (Experimental): Benzathine Penicillin G treatment
  Interventions: Drug: Benzathine Penicillin G
- Molecular subtyping (others) of Treponema pallidum (Experimental): Benzathine Penicillin G treatment
  Interventions: Drug: Benzathine Penicillin G

INTERVENTIONS:
Drug: Benzathine Penicillin G

SUMMARY:
The investigators compare the treatment results and clicical presentations of different Molecular subtyping of Treponema pallidum

ELIGIBILITY:
Inclusion Criteria

1. Persons with confirmed early symptomatic syphilis (primary or secondary) or high-titer latent syphilis

Exclusion Criteria:

1. Pregnant woman
2. Known allergy to penicillin
3. RPR titers were found to be 1:8 or less

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-08; Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
rapid plasma regain titer | 6 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology and Venereology, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China, Beijing, China